CLINICAL TRIAL: NCT05962203
Title: SHIP-AGE: Frailty, Renal Function, and Multi-component Primary Care in Rural Mecklenburg-Western Pomerania.
Acronym: MV-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BB 161/22
Record Dates: First submitted 2023-06-13; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Frailty Syndrome
Keywords: Chronic kidney disease; Frailty; Falls; Cognitive decline; Multi-component interventions; Rural communities
MeSH Terms: conditions — Frailty; Renal Insufficiency, Chronic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Multivariable logistic regression; Multivariable Cox regression, Chi-Square-Test, Propensity score matching
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-factorial geriatric assessment, monitoring & management systems (Experimental): All participants in the observational/interventional study (MV-FIT) will receive guideline-based, multi-factorial geriatric assessment, monitoring & managements (multi-component healthcare). Other: GFR Measuremments, Blood sampling, Urine sampling
  Interventions: Diagnostic Test: Multi-factorial geriatric assessment, monitoring & management systems

INTERVENTIONS:
Diagnostic Test: Multi-factorial geriatric assessment, monitoring & management systems — Multi-factorial geriatric assessment, monitoring & management systems, e.g. community-based and home-based exercise programs, polypharmacy
  Other Names: Community-based and home-based exercise programs

SUMMARY:
Chronic kidney disease (CKD) is a leading risk factor for cardiovascular and all-cause mortality among the elderly. Mecklenburg-Western Pomerania has the largest prevalence of CKD in Germany and Europe. The CKD impact in primary care strategies to reduce frailty syndrome in the elderly is unknown. For this purpose, about 820 elderly participants will be included in an observational study (MV-FIT), who will undergo an multi-factorial geriatric assessment, monitoring & management program, specifically designed to avoid frailty. The goal of the full-scale study is to evaluate the impact of CKD in multi-component primary care strategies to reduce frailty among elderly persons in rural Mecklenburg-Western Pomerania. MV-FIT will be conducted on individuals in rural Mecklenburg-Western Pomerania, who will be observed over a period of 3 years. The Study of Health in Pomerania (SHIP) is a population-based epidemiological, two independent-cohort, study (SHIP and SHIP-TREND). SHIP cohorts have been followed for >24 years. SHIP/SHIP TEND participants >60 years or older will studied by a follow-up survey. The aim is to gain new insights into the development of frailty and to develop strategies for keeping those affected healthy.

DETAILED DESCRIPTION:
Our study is a longitudinal population-based epidemiological SHIP-cohort study combined with a prospective, multi-centered, observational/interventional investigation. MV-FIT is an observational study of individuals aged 65 years or older with mGFR >30 mL/min (n=~820). All participants in the observational/interventional study will receive guideline-based, multi-factorial geriatric assessment, monitoring & managements (multi-component healthcare). Subjects will be stratified by mGFR. Objectives are 1) to implement multi-component healthcare specifically comprised of components to reduce frailty and incident falls, 2) to improve compliance and adherence to the multi-component healthcare for frailty and improvement of patient welfare, ability to live independently, quality-of-life, number of falls, referrals to nursing homes, all-cause mortality in primary care of the elderly, 3) to seek the elderly individuals' experience during the course of multi-factorial primary care intervention through In-depth interviews, 4) to clarify the burden of CKD on frailty and health status, and 5) to identify novel risk factors and mechanisms for frailty and pre-frailty. MV-FIT data will be corroborated by SHIP/SHIP-TREND data.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* mGFR > 30 mL/min per 1.73 m2
* being able to understand and give written informed consent.

Exclusion Criteria:

* bedridden
* palliative
* inability to consent
* severe dementia
* inability to speak
* lack of compliance (paracusis, inability to fulfill at least 60% of the assessments)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Frailty | from baseline to follow-up at 36 month
  The primary outcome will be frailty from baseline to follow-up at 36 months post subject inclusion (i.e. Frail vs. non-Frail). The frailty phenotype defines frailty as a clinical syndrome meeting three or more of five phenotypic criteria: (1) unintentional body weight loss (2) slow walking pace, (3) self-reported exhaustion, (4) muscle weakness, and (5) self-reported low physical activity.
body weight loss | 36 months
  unintentional body weight loss (determined weight in kilograms); see phenotype criteria (# 1) above
slow walking pace | 36 months
  slow walking pace (determined by walking speed measurements in m/sec); see phenotype criteria (# 2) above
exhaustion | 36 months
  self-reported exhaustion (determined by questionnaire), see phenotype criteria (# 3) above
muscle weakness | 36 months
  muscle weakness (determined by handgrip and jump strengths in kg); see phenotype criteria (# 4) above
low physical activity | 36 months
  (5) self-reported low physical activity (determinded by questionnaire); see phenotype criteria (# 5) above

SECONDARY OUTCOMES:
Frailty transition | 36 months
  Frailty transition (pre-frailty, in which one or two criteria (see above) are present)
mGFR transition | 36 months
  mGFR transition (transition from GFR KDIGO (Kidney Disease: Improving Global Outcomes) Stage 2 CKD in mL/min per 1.73 m2 to KDIGO Stage 3 in mL/min per 1.73 m2)
patient welfare | 36 months
  self-reported patient welfare (questionnaire)
ability to live independently | 36 months
  self-reported ability to live independently (Barthel Index for Activities of Daily Living (ADL))
cognitive decline | 36 months
  cognitive decline
number of falls | 36 months
  self-reported number of falls
admission to hospitals | 36 months
  self-reported admission to hospitals
referrals to nursing homes | 36 months
  self-reported referrals to nursing homes
mortality | 36 months
  all-cause mortality in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Maik Gollasch, MD, PhD, Principal Investigator — University Medicine Greifswald

IPD SHARING:
Plan to Share IPD: No